CLINICAL TRIAL: NCT02567539
Title: Phase II Study of Hypofractionated Stereotactic Radiotherapy for Patients With Recurrent High Grade Glioma
Brief Title: Hypofractionated Stereotactic Radiotherapy for Patients With Recurrent High Grade Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1394
Record Dates: First submitted 2015-09-28; First posted 2015-10-05 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Recurrent High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recurrent high grade glioma (Experimental): IMRT with or without radiosensitive therapy
  Interventions: Radiation: IMRT with or without radiosensitive therapy; Drug: Radiosensitive therapy

INTERVENTIONS:
Radiation: IMRT with or without radiosensitive therapy — Re-irradiation with hypofractionated intensity modulated radiation therapy (IMRT), using VMAT RapidArc
  Other Names: Hypofractionated Stereotactic Radiation
Drug: Radiosensitive therapy — Radiosensitive therapy with Temozolomide
  Other Names: Chemotherapy

SUMMARY:
The study is aimed to evaluate efficacy and safety of re-irradiation for patients with recurrent high grade gliomas after other treatment.

DETAILED DESCRIPTION:
Investigators designed this study of a re-irradiation with single radiosurgery or hypofractionated intensity modulated radiation therapy (IMRT) with or without temozolomide.

Objective of the study is evaluating efficacy and safety of re-irradiation for patients with recurrent high grade gliomas after other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Karnosky performance status (KPS) ≥70
* Patients aged >70 years with KPS ≥80
* Histopathologically confirmed grade III-IV glioma
* Estimated survival ≥ 3 months
* Any Tumor volume
* Unifocal tumor
* Interval time from previous radiotherapy ≥ 6mesi
* Normal liver, Kidney and bone marrow function
* Written informed consent

Exclusion Criteria:

* KPS < 70
* Multifocal tumor
* Other primary cancer
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Progression free of participants | 4 years
Overall survival of participants | 4 years

SECONDARY OUTCOMES:
Incidence of radionecrosis | 3 months
Questionnaire assessment of neurocognitive function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Piera Navarria, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Result] Navarria P, Ascolese AM, Tomatis S, Reggiori G, Clerici E, Villa E, Maggi G, Bello L, Pessina F, Cozzi L, Scorsetti M. Hypofractionated Stereotactic Radiation Therapy in Recurrent High-Grade Glioma: A New Challenge. Cancer Res Treat. 2016 Jan;48(1):37-44. doi: 10.4143/crt.2014.259. Epub 2015 Feb 23. PMID 25761491
- [Result] Scorsetti M, Navarria P, Pessina F, Ascolese AM, D'Agostino G, Tomatis S, De Rose F, Villa E, Maggi G, Simonelli M, Clerici E, Soffietti R, Santoro A, Cozzi L, Bello L. Multimodality therapy approaches, local and systemic treatment, compared with chemotherapy alone in recurrent glioblastoma. BMC Cancer. 2015 Jun 30;15:486. doi: 10.1186/s12885-015-1488-2. PMID 26118437
- [Derived] Navarria P, Pessina F, Clerici E, Bellu L, Franzese C, Franzini A, Simonelli M, Bello L, Santoro A, Politi LS, D'agostino GR, Casarotti A, Fernandes B, Torri V, Scorsetti M. Re-irradiation for recurrent high grade glioma (HGG) patients: Results of a single arm prospective phase 2 study. Radiother Oncol. 2022 Feb;167:89-96. doi: 10.1016/j.radonc.2021.12.019. Epub 2021 Dec 22. PMID 34952000